CLINICAL TRIAL: NCT02702063
Title: Calibrating Cardiac Output Measurement of Electrical Cardiometry With Transthoracic Echocardiography
Acronym: EC vs TTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Clemens Ortner, Assistant Professor, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MUVienna 1139/2015
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TTE vs. EC + calibration group (Other): 50 Patients undergoing routine transthoracic echocardiography at laboratory for transthoracic echocardiography at the department of cardiology of Medical University Vienna will be enrolled following informed consent. Non-inclusion criteria are inability to understand study procedure and age under 18 years old.
  Patients with any grade of aortic regurgitation, congenital heart disease with intracardiac shunt (left-right shunt or right-left shunt) or arrhythmia (atrial fibrillation) or withdrawing consent during study procedure will be excluded. In addition, patients with intraabdominal (IAH), intracranial (ICH) hypertension or any disease of the hip joint, will not be included into the trial.
  Interventions: Other: TTE vs. EC + calibration group
- Right heart catheterisation (Other): Twenty five patients undergoing routine right heart catheterization (RHC) at the department of cardiology for the evaluation of suspected pulmonary hypertension or heart failure will be included in this trial. EC measurements will be obtained during RHC, and a TTE (for measuring LVOT-area) will be performed immediately before undergoing RHC. Inclusion and exclusion criteria are similar as described above.
  Interventions: Procedure: right heart catheterisation
- Passive leg raising test (Other): 50 Patients undergoing routine transthoracic echocardiography at laboratory for transthoracic echocardiography at the department of cardiology of Medical University Vienna will be enrolled following informed consent. Non-inclusion criteria are inability to understand study procedure and age under 18 years old.
  Patients with any grade of aortic regurgitation, congenital heart disease with intracardiac shunt (left-right shunt or right-left shunt) or arrhythmia (atrial fibrillation) or withdrawing consent during study procedure will be excluded. In addition, patients with intraabdominal (IAH), intracranial (ICH) hypertension or any disease of the hip joint, will not be included into the trial.
  SV and CO will be measured using TTE and EC. Patient's legs will then be raised by 45degree, and SV and CO measurements will be repeated after 1 minute. Changes in SV and CO observed with both methods will be compared.
  Interventions: Other: passive leg raising test

INTERVENTIONS:
Other: passive leg raising test — Patients undergoing routine echocardiography are exposed to a passive leg raising test. Change in SV will be measured by TTE and compared to changes in SV measured by EC.
  Arms: Passive leg raising test
Procedure: right heart catheterisation — CO in patients undergoing routine right heart catheterisation will be measured and compared between 3 methodologies: right heart catheterisation, TTE and EC
  Arms: Right heart catheterisation
Other: TTE vs. EC + calibration group — Patients will undergo routine echocardiography. CO and SV will be measured by TTE and compared to measurements obtained from simultaneous EC-measurements.
  Arms: TTE vs. EC + calibration group

SUMMARY:
Cardiac output (CO) is a key variable when describing the cardiovascular system. Electrical cardiometry (EC) is a non-invasive method in measuring stroke volume and cardiac output. However, its accuracy has been inconsistent. Therefore Martin et al. have compared measurements with echocardiographic measurements and propose calibration with left ventricle outflow tract (LVOT)-measurements obtained from transthoracic echocardiography (TTE). This study was performed in pregnant women at term. Goal of this study is to validate their formula in non-pregnant outpatients undergoing echocardiography for cardiology work-up. Secondary aim is to perform a leg raising test and to compare changes in stroke volume observed with either EC or TTE.

DETAILED DESCRIPTION:
Cardiac output (CO) is a key variable when describing and treating the cardiovascular system. The ideal cardiac output (CO) monitor would be safe, non-invasive, low-cost, painless, easy to interpret and would allow for the continuous, hands-free acquisition of accurate data. Electrical cardiometry (EC), a more recent version of impedance cardiography (ICG), meets many of the criteria for an ideal monitor and previously published research suggests that EC successfully trends CO1-3, but its accuracy in measuring absolute values of stroke volume (SV) has been inconsistent in published research4-8. Electrical cardiometry works by sending an insensible high frequency alternating current through the thorax and measures changes in thoracic impedance that are attributed to systolic blood flow acceleration over the cardiac cycle. Using fiducial points in the tracing of the first derivative of impedance, EC calculates left ventricular ejection time (LVET) and mean velocity of blood during systole. By further estimating a patient constant that is primarily based on body mass ('volume of electrically participating tissue' (VEPT)), stroke volume is estimated in the following way:

- SVEC = VEPT * Mean blood velocity * corrected Flow Time (FTc).

Cardiac output monitors are typically validated against a reference standard, which has traditionally been thermodilution using a pulmonary artery catheter (PAC). Given the risks associated with the use of pulmonary artery catheters9 an alternative method, such as transthoracic echocardiography (TTE), lends itself as valuable substitute technique for measuring CO. Transthoracic echocardiography is safe, painless and non-invasive. Similarly to EC, SV estimate by TTE is based on a measurement of mean blood velocity and ejection time (mean blood velocity x ejection time = velocity time integral, VTI; (Figure 3)). However, in contrast to EC, the parameters for blood velocity and left ventricular ejection time are not multiplied with a normative patient constant, but with a measured parameter: the left ventricular outflow tract area (LVOT area):

- SVTTE = LVOT area * mean blood velocity * ejection time. Main disadvantage of using TTE for CO-measurement is advanced training that is needed to obtain VTI measurements and that it is highly labor intense to obtain repeated VTIs for continuous or repeated CO measurements. Measurement of LVOT area, by contrast, is a one-time measurement obtained from parasternal long axis view, which necessitates only basic training of TTE.

Recently Martin and colleagues10 compared SV parameters derived from EC and TTE in a sample of 44 healthy pregnant volunteers and found excellent agreement in mean left ventricular ejection time and heart rate. However, agreement in SV was poor with a percentage error of 42% in Bland-Altman analysis. Hypothesizing that both methodologies in estimating SV, EC and TTE, use measures for blood velocity and systolic ejection time, Martin et al. hypothesized that agreement between both methods could be significantly improved by calibrating SV-EC with the LVOT area that is derived from one time TTE measurement. Based on a multiplicative linear regression model and following log-linear transformation Martin et al. derived the following formula for calibration:

SVEC_Modified = 2.2 * LVOT_area(0.705) * SV_EC(0.388) * Weight(0.21) By applying this formula, agreement in SV measurements significantly improved and percentage error decreased to 22 %. However, data was derived from a very specific patient population (pregnant women) and accuracy of the modified SV-assessment was not validated in a prospective manner.

Therefore, this study proposes to compare SV-estimates derived from EC and TTE in non-pregnant outpatients undergoing routine echocardiography assessment. Primary aim of this study is to evaluate if agreement between both methods can be improved by calibrating SV-measurements obtained from electrocardiometry with a one-time LVOT area measurement obtained from TTE.

Secondary aim will be to perform passive leg raising test and compare sensitivity in both identifying fluid responsiveness between both monitoring methodologies.

Third aim is to compare CO derived measurements from EC and TTE with gold standard measurements derived from patients undergoing routine right heart catheterisation for evaluation of cardiac and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* able to understand study procedure

Exclusion Criteria:

* aortic regurgitation
* congenital heart disease with intracardiac shunt
* arrhythmia
* withdrawing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
agreement Stroke volume | 3 seconds
  SV measured by TTE, RHC and EC will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No